CLINICAL TRIAL: NCT06006858
Title: Safety Profile Following Moderna COVID-19 Primary Vaccine in Healthy Adults Aged ≥ 18 Years in Indonesia
Brief Title: Post Authorization Safety Study Moderna COVID-19 Primary Vaccine
Status: Completed | Type: Observational
Sponsor: PT Bio Farma (Industry)
Collaborators: National Advisory Immunization Committee Indonesia (Unknown)
Responsible Party: Sponsor
Other Study IDs: COV19M-0422
Record Dates: First submitted 2023-08-22; First posted 2023-08-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: COVID-19; Moderna Vaccine; Safety Vaccine
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderna COVID-19 Vaccine: Clinically healthy adults aged ≥ 18 years who received Primary Moderna COVID-19 Vaccine
  Interventions: Biological: Moderna COVID-19 Vaccine

INTERVENTIONS:
Biological: Moderna COVID-19 Vaccine — Moderna COVID-19 Vaccine is provided as a white to off-white suspension for intramuscular injection. Each 0.5 mL dose of Moderna COVID-19 Vaccine contains 100 mcg of nucleoside-modified messenger RNA (mRNA) encoding the pre-fusion stabilized Spike glycoprotein (S) of SARS-CoV-2 virus.

SUMMARY:
This study is Post Authorization Safety Study (PASS) Phase IV of Moderna COVID-19 Primary Vaccine

DETAILED DESCRIPTION:
This study is Post Authorization Safety Study (PASS) Phase IV, to assess any local and systemic reaction after immunization with Moderna COVID-19 vaccine using retrospective cohort study trial design to assess safety profile following Moderna COVID-19 primary vaccine in healthy adults aged ≥ 18 years in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy adults aged ≥ 18 years.
* Subjects have been informed properly regarding the study and accepted to be enrolled in this study.

Exclusion Criteria:

- Subjects concomitantly enrolled or scheduled to be enrolled in another trial at the time of receiving the Moderna COVID-19 vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged ≥ 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1284 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Local Reactions Following Moderna COVID-19 Vaccine | 28 Days after each dose
  Percentage of subject with local reactions following immunization with Moderna COVID-19 vaccine.
Systemic Reactions Following Moderna COVID-19 Vaccine | 28 Days after each dose
  Percentage of subject with systemic reactions following immunization with Moderna COVID-19

SECONDARY OUTCOMES:
Immediate Reactions | 30 minutes after each dose
  percentage of subject with adverse event following immunization with Moderna COVID-19 vaccine.
1-3 Days Reactions | 1-3 minutes after each dose
  percentage of subject with adverse event following immunization with Moderna COVID-19 vaccine.
4-7 Days Reactions | 4-7 Days after each dose
  percentage of subject with adverse event following immunization with Moderna COVID-19 vaccine.
8-28 Days Reactions | 8-28 Days after each dose
  percentage of subject with adverse event following immunization with Moderna COVID-19 vaccine.
Serious Reactions | 28 Days after each dose
  Any serious adverse events following immunization with Moderna COVID-19 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Julitasari Sundoro, MD, Principal Investigator — National Advisory Immunization Committee
Locations (18):
- Indonesia (18):
  - Gambir Public Health Center, Jakarta Pusat, Jakarta Special Capital Region
  - Johar Baru Public Health Center, Jakarta Pusat, Jakarta Special Capital Region
  - Cempaka Putih Public Health Center, Jakarta Pusat, Jakarta Special Capital Region
  - Kemayoran Public Health Center, Jakarta Pusat, Jakarta Special Capital Region
  - Palmerah Public Health Center, Jakarta
  - Kebon Jeruk Public Health Center, Jakarta
  - Cengkareng Public Health Center, Jakarta
  - Kebayoran Lama Public Health Center, Jakarta
  - Tebet Public Health Center, Jakarta
  - Setiabudi Public Health Center, Jakarta
  - Pulo Gadung Public Health Center, Jakarta
  - Duren Sawit Public Health Center, Jakarta
  - Regional Hospital Duren Sawit, Jakarta
  - Kramat Jati Public Health Center, Jakarta
  - Cilincing Public Health Center, Jakarta
  - Koja Public Health Center, Jakarta
  - Tanjung Priok Public Health Center, Jakarta
  - Pademangan Public Health Center, Jakarta

IPD SHARING:
Plan to Share IPD: No